CLINICAL TRIAL: NCT06537011
Title: An Exploratory Phase II Study of Neoadjuvant Treatment With AK112 Plus AP Regimen for Operable Locally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: AK112 Plus AP Regimen for Operable Locally Advanced Head and Neck Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK112-II-020
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Neoadjuvant Therapy of Operable Locally Advanced Head and Neck Squamous Cell Carcinoma
Keywords: neoadjuvant therapy,AK112,advanced head and neck squamous cell carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK112 combined with AP neoadjuvant therapy (Experimental): Three cycles of AK112 were given before operation every 3 weeks on D 1, D 22 and D 43, while AP regimen was given every 3 weeks on D 1, D 22 and D 43, respectively.
  Interventions: Drug: AK112

INTERVENTIONS:
Drug: AK112 — 1. The patients are given AK112 combined with AP regimen every 3 weeks for 3 cycles before operation.
  2. After the neoadjuvant therapy ,the patients will be assessed and be commanded surgery.
  3.4-6 weeks after the surgery, the patients will be given chemoradiotherapy or radiotherapy alone decided on the conditon after surgery.
  4.The participants will receive AK112 for 14 cycles after surgery.

SUMMARY:
This exploratory phase II study is designed to enroll patients with operable locally advanced head and neck squamous cell carcinoma, to observe the efficacy and safety of AK112 combined with chemotherapy as neoadjuvant therapy on them.

DETAILED DESCRIPTION:
This exploratory phase II study is designed to enroll 36 patients with operable locally advanced head and neck squamous cell carcinoma(defined according to 8th teh edition of AJCC Guideline). The patients are given 3cycles of AK112(20mg/Kg per cycle) combined with AP regimen(platinum based chemotherapy), with a 3-week interval between each cycle (d1,d22,d43). After 3 cycles' therapy, if the volume of primary tumor decreases by over 50%，the range of resection operation will be conducted by the actual range of tumor, or else the surgery will be conducted by the original range of the tumor. The adjuvant radiation therapy would be conducted in 4-6 weeks after the surgery, while the adjuvant therapy of AK112 would be given in 21days after the surgery for 14 cycles. The process will continue until disease progression or uncontrolled toxicity. The primary endpoint is pCR(pathological complete response) and 2y-EFS; the secondary endpoint is MPR(Main pathological response)、ORR(objective response rate)、2y-OS(overall survival)、organ retention rate and safety assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years, regardless of sex;
2. histological diagnosis of squamous cell carcinoma in oral cavity,oropharynx, hypopharynx or laryngeal;
3. preoperative evaluation turns to be operatable;
4. locally advanced, according to the American Joint Committee on Cancer ( AJCC -RSB- guidelines, 8th edition),HPV status is determined by p16 immunohistochemistry (IHC);
5. Have not received prior treatment for head and neck squamous cell carcinoma;
6. Have at least one evaluable target lesion according to RECIST version 1.1;
7. ECOG physical condition 0-1 point;
8. The function of the major organs is normal, which meets the following criteria(not receiving blood transfusion in 14 days):

   a. Hb(hemoglobin)≥90g/L:b. ANC(Neutrophils)≥1.5x109/L; c. PLT(platelet)≥80x109／L；

   The biochemical tests should meet the following criteria:

   a.BIL(bilirubin)< 1.25 times the upper limit of normal (ULN); b.ALT(Alanine aminotransferase) and AST(Aspartate aminotransferase)<2.5xULN; c.Serum CR(creatinine) ≤ ULN, endogenous creatinine clearance > 50 ml/min (Cockcroft-Gaut formula) ;
9. Sign a written informed consent form before performing any test related activities;
10. The researchers judged that they were able to comply with the study protocol;
11. Pregnancy test (for fertile women) was negative at screening;
12. Fertile male patients as well as fertile female patients at risk of fertility and pregnancy had to agree to use 2 contraceptive methods throughout the study period (at least one of which was considered to be an efficient contraceptive method) .
13. Patients who are willing and able to follow visiting schedules, treatment plans, laboratory tests, and other research procedures.

Exclusion Criteria:

1. Previously received immunotherapy with anti-PD-1(programmed cell death receptor-1), anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibodies (including ipilimumab) or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways;
2. Previously received prior chemotherapy or antiangiogenic therapy;
3. Received major surgery ≤4 weeks before admission;
4. Carrying any active autoimmune disease or history of autoimmune disease'
5. Previous or concurrent getting cancers (except those that have been cured and have survived cancer-free for more than 5 years, such as skin basal-cell carcinoma, cervical carcinoma in situ, and papillary thyroid cancer) .
6. Uncontrollable clinical symptom or disease of the heart;
7. Within 14 days before the administration of the study drug, subjects who were required to undergo systemic therapy with corticosteroid (> 10 mg daily prednisone efficacy dose) or other immunosuppressive agents, in the absence of active autoimmune disease, adrenal hormone replacement with inhaled or topical steroids and a therapeutic dose of prednisone > 10 mg/day was allowed;
8. Active infection requiring treatment;
9. Patients with congenital or acquired immunodeficiency(such as HIV),active hepatitis B (HBV-DNA ≥104 copies/ml or 2000 IU/ml) , or hepatitis C (HCV-RNA was above the lower limit of detection);
10. The patient has received other cancer specialised treatment;
11. The live vaccine was administered within 4 weeks before starting the study;
12. Known history of psychotropic substance abuse, alcohol or drug abuse;
13. Pregnant or lactating female;
14. The researchers determined that the subjects had other factors that could have led them to stop the study mid-course, such as having a serious medical condition (including mental illness) that required combined treatment, and severe abnormalities in laboratory tests, family or social factors that may affect the safety of the subject or the collection of experimental data;
15. A patient who is considered by the surgeon to be inoperable;
16. Active tuberculosis;
17. Severe infections (including, but not limited to, hospitalizations for infections, bacteremia, or complications of severe pneumonia) occurring within 4 weeks before study initiation;
18. Received systemic immunostimulatory medication (including but not limited to interferon or interleukin-2[ IL-2]) within 4 weeks before initiation of study treatment or remained within 5 drug half-lives (taking the older of the two) .

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2027-07-15 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
EFS | 2 years
  The time between the onset of treatment till disease progression, discontinuation of treatment for any reason, or death

SECONDARY OUTCOMES:
pCR | 3 cycles of treatment(1.5months)
  The percentage of tumor tissue that has completely disappeared on pathological examination after treatment
OS | 2 years
  The time between the onset of treatment till death
MPR | 3 cycles of treatment(1.5months)
  The percentage of active tumor components decreasing below a certain threshold

IPD SHARING:
Plan to Share IPD: No